CLINICAL TRIAL: NCT01799720
Title: Effect of Omega-3 Dietary Supplements With Different Oxidation Levels in the Lipidic Profile of Women: a Randomized Controlled Trial
Brief Title: Oxidized Omega-3 Supplements With Different Oxidation
Acronym: GPTPASPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); University of Alicante (Other)
Responsible Party: Principal Investigator, Elena García García, PhD,PID, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Elena García-García; Enrique Roche Collado (Other Grant/Funding Number: Instituto de Salud Carlos III-FEDER PS09/01093); Vicente Micol Molina (Other Grant/Funding Number: PROMETEO/2012/007 from Generalitat Valenciana); Enrique Roche Collado (Other Grant/Funding Number: CIBERobn (CB12/03/30038))
Record Dates: First submitted 2013-02-19; First posted 2013-02-27 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Overweight
Keywords: blood cholesterol; blood lipid profile; triglycerides; commercial pills; fish oil; lipid peroxidation; Circulating lipidic profile
MeSH Terms: conditions — Overweight | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Less oxidized oil and diet (Experimental): Analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose we have designed a single-blind, parallel-groups, randomized controlled trial. Participants from group 1 took 2 capsules/day of one of the less oxidized oil (containing 300 mg EPA + DHA) and diet. Follow-up 30 days
  Interventions: Dietary Supplement: Less oxidized oil and diet
- More oxidized oil and diet (Experimental): Analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose we have designed a single-blind, parallel-groups, randomized controlled trial. Participants from group 2 took 2 capsules/day of one of the most oxidized oil (containing 300 mg EPA + DHA) and diet . Follow-up 30 days
  Interventions: Dietary Supplement: More oxidized oil and diet
- Hypercholesterolemic diet (Experimental): Analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose we have designed a single-blind, parallel-groups, randomized controlled trial. Participants from group 3 only took diet and no capsules. Follow-up 30 days
  Interventions: Drug: Hypercholesterolemic diet

INTERVENTIONS:
Dietary Supplement: Less oxidized oil and diet — Analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose we have designed a single-blind, parallel-groups, randomized controlled trial. Finally 52 women between 25 and 75 years old randomly were distributed into three groups. Participants from group 1 took 2 capsules/day of one of the less oxidized oil (containing 300 mg EPA + DHA) and diet, . Follow-up 30 days
  Other Names: less oxidized oil
  Arms: Less oxidized oil and diet
Dietary Supplement: More oxidized oil and diet — Analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose we have designed a single-blind, parallel-groups, randomized controlled trial. Finally 52 women between 25 and 75 years old randomly were distributed into three groups. Participants from group 2 took 2 capsules/day of one of the more oxidized oil (containing 300 mg EPA + DHA) and diet . Follow-up 30 days
  Other Names: More oxidized oil
  Arms: More oxidized oil and diet
Drug: Hypercholesterolemic diet — Analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose we have designed a single-blind, parallel-groups, randomized controlled trial. Finally 52 women between 25 and 75 years old randomly were distributed into three groups. Participants from group 3 only received the diet and no capsules. Follow-up 30 days
  Arms: Hypercholesterolemic diet

SUMMARY:
The oxidation level of unsaturated fatty acid supplements commercialized in capsules could be a serious problem for manufacturers and a risk to consumers; health by ingesting substances whose effects are not desired. Therefore, the main objective of this paper is to analyze the effect of dietary supplements Omega-3 with different levels of oxidation in the lipid profile of women who consume these supplements. For this purpose the investigators have designed a single-blind, parallel-groups, randomized controlled trial. Finally, 52 women between 25 and 75 years old were randomly distributed into three groups: (1) took 2 capsules/day of one of the less oxidized oil (containing 300 mg EPA + DHA) and diet, (2) took 2 capsules/day of one of the most oxidized oil (containing 300 mg EPA + DHA) and diet and (3) no capsules, only received the diet. There was a 30 days follow-up . All groups followed a low cholesterol diet. Circulating glucose, total cholesterol, triglycerides and glutamic pyruvic transaminase were determined at the beginning and end of a 30 day period.

DETAILED DESCRIPTION:
The assignment of women to distinct groups was carried out following the classification criteria established by (NCEP, 2002), and performed by the research team. Women were randomly assigned to one of three parallel groups, in a near 1:1:1 ratio. Group 1 (n=20) took two capsules per day of less oxidized oil (containing 300 mg EPA-DHA per capsule) and diet. Group 2 (n=18) consumed two capsules per day of oxidized oil (containing 300 mg EPA-DHA per capsule) and diet. Finally, group 3 (n=19) performed the diet but did not take any capsule. Therefore, the design was a single-blind (participants did not know what type of capsule they were receiving), parallel-group, randomized controlled trial conducted at the Miguel Hernández University of Elche (Spain).

Statistical analysis was carried out using STATGRAPHICS Centurion XV software (StatPoint Technologies, Inc. Warrington, VA); likewise, significance was defined at p<0.05. Data are reported as mean standard error of the mean (SEM). Intragroup statistical comparisons were performed using the following hypothesis tests, both parametric and non-parametric: t-test, sign test and signed rank test for paired samples. Intergroup statistical comparisons were performed using the one-way analysis of variance (ANOVA) and the Kruskal-Wallis hypothesis tests. Also, Fisher least significant difference (LSD)Multiple Range Test and Tukey HSD were used in order to determine which means were significantly different from the others.

Methods for additional analyses Generalized multiple regression was used to statistically analyse the relationships between the variations in the lipid profile and the consumption of w-3 dietary supplements.

ELIGIBILITY:
Inclusion Criteria:

* presence of dyslipemia with no indication of drug treatment
* blood cholesterol levels ranging 250-300 mg/dL
* triglycerides (TG) 160-175 mg/dL

Exclusion Criteria:

* pregnancy
* lactation
* participation in another supplementary feeding programme

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena García, PDI, Principal Investigator — Universidad Miguel Hernandez de Elche
Locations (1):
- Pharmacy Iborra Campos, Elche, Alicante, Spain

REFERENCES:
- [Derived] Garcia-Hernandez VM, Gallar M, Sanchez-Soriano J, Micol V, Roche E, Garcia-Garcia E. Effect of omega-3 dietary supplements with different oxidation levels in the lipidic profile of women: a randomized controlled trial. Int J Food Sci Nutr. 2013 Dec;64(8):993-1000. doi: 10.3109/09637486.2013.812619. Epub 2013 Jul 18. PMID 23863036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The place where women were recruited for our study was a pharmacy located in the city centre of Elche, during October 2010. Elche is an industrial city located in the Southeast of Spain, with a population of 230 000 inhabitants.
Pre-assignment Details: Before the survey began, 14 people were discarded from the survey because their cholesterol levels were lower than the inclusion standards.
  5 participants decided to withdraw from the survey once it had began. 3 of them abandoned the study voluntarily. 1 left because she was pregnant, and 1 violated the protocol norms and was expelled.
Groups:
- Less Oxidized Oil and Diet: Participants from group 1 took 2 capsules a day of one of the less oxidized oil (containing 300 mg EPA + DHA) and diet, Follow-up 30 days
- More Oxidized Oil and Diet: Participants from group 2 took 2 capsules a day of one of the more oxidized oil (containing 300 mg EPA + DHA) and diet, Follow-up 30 days
- Diet: Participants from group 3 took only diet, Follow-up 30 days
Period: Overall Study
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Started | 20 | 18 | 19
Began the Treatment | 20 | 18 | 19
Began the Treatment and Finished it | 17 | 17 | 18
Completed | 17 | 17 | 18
Not Completed | 3 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Less Oxidized Oil and Diet: Participants from group 1 took 2 capsules/day of one of the less oxidized oil (containing 300 mg EPA + DHA) and diet. Follow-up 30 days.
- More Oxidized Oil and Diet: Participants from group 2 took 2 capsules/day of one of the most oxidized oil (containing 300 mg EPA + DHA) and diet. Follow-up 30 days.
- Only Diet: Participants from group 3 only received the diet. Follow-up 30 days.
- Total: Total of all reporting groups
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Only Diet | Total
Number analyzed (Participants) | 17 | 17 | 18 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 14 | 41
  >=65 years | 3 | 4 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.65 (12.65) | 56.82 (12.18) | 51.94 (10.80) | 55.14 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 18 | 52
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 17 | 17 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Weight (Kilogram) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30)
Description: In this table the investigators present the weight (kilogram) of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: kilogram
Groups:
- More Oxidized Oil and Diet: Participants from group 2 took 2 capsules/day of one of the more oxidized oil (containing 300 mg EPA + DHA) and diet. Follow-up 30 days.
- Diet: Participants from group 3 only took diet. Follow-up 30 days.
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
kilogram
  Day 1 | 70.17 (3.71) | 68.77 (3.42) | 75.15 (3.95)
  Day 30 | 69.38 (3.61) | 67.78 (3.41) | 74.29 (3.94)

2. Secondary Outcome: Height (Metre) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the height of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: metres
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
metres
  Day 1 | 1.60 (0.02) | 1.59 (0.01) | 1.61 (0.01)
  Day 30 | 1.60 (0.02) | 1.59 (0.01) | 1.61 (0.01)

3. Secondary Outcome: Body Mass Index (BMI) (Kg/m2) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the Body Mass Index of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: kilogram / square metre
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
kilogram / square metre
  Day 1 | 27.43 (1.41) | 28.65 (2.13) | 29.00 (1.50)
  Day 30 | 27.10 (1.34) | 26.94 (1.36) | 28.64 (1.45)

4. Secondary Outcome: Hip/Waist Ratio of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30)
Description: In this table the investigators present the hip/waist ratio of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: ratio*100
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
ratio*100
  Day 1 | 86.5 (2.1) | 87.2 (3.0) | 86.0 (2.9)
  Day 30 | 86.5 (2.1) | 87.2 (3.0) | 86.0 (2.9)

5. Secondary Outcome: Systolic Pressure (mmHg) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the systolic pressure of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: millimetres of mercury
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
millimetres of mercury
  Day 1 | 129.9 (0.50) | 123.7 (0.66) | 118.6 (0.37)
  Day 30 | 118.2 (0.42) | 120.2 (0.41) | 119.4 (0.41)

6. Secondary Outcome: Diastolic Pressure (mmHg) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the diastolic pressure of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: millimetres of mercury
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
millimetres of mercury
  Day 1 | 77.2 (0.26) | 73.9 (0.34) | 73.3 (0.34)
  Day 30 | 68.9 (0.21) | 75.1 (0.29) | 72.8 (0.20)

7. Secondary Outcome: Glucose (mg/dL) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the glucose of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: milligram / decilitre
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
milligram / decilitre
  Day 1 | 103.35 (3.18) | 108.96 (11.11) | 99.72 (4.53)
  Day 30 | 116.24 (4.30) | 111.37 (2.46) | 108.26 (2.55)

8. Secondary Outcome: Cholesterol (mg/dL) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the cholesterol of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: milligram / decilitre
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
milligram / decilitre
  Day 1 | 246.64 (12.92) | 232.94 (12.55) | 236.78 (4.17)
  Day 30 | 217.76 (8.98) | 237.52 (7.54) | 227.22 (6.02)

9. Secondary Outcome: Triglycerides (TGs) (mg/dL) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the Triglycerides (TGs) of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: milligram / decilitre
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
milligram / decilitre
  Day 1 | 164.41 (15.43) | 160.41 (11.34) | 174.83 (19.83)
  Day 30 | 125.52 (12.34) | 116.88 (11.43) | 130.04 (10.18)

10. Secondary Outcome: Glutamic Pyruvic Transaminase (GPT) (U/L) of Volunteers at the Beginning (Day 1) and at the End of the Study (Day 30).
Description: In this table the investigators present the Glutamic Pyruvic Transaminase (GPT) of the three intervented groups. Data are mean ± sem.
Time Frame: Days 1 and 30
Measure: Mean (Standard Error); unit: Units / litre
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Number analyzed (Participants) | 17 | 17 | 18
Units / litre
  Day 1 | 22.70 (2.71) | 24.90 (2.96) | 23.54 (3.92)
  Day 30 | 20.69 (3.34) | 18.46 (1.62) | 19.94 (2.19)

ADVERSE EVENTS:
Description: 5 participants decided to withdraw from the survey once it had began. 3 of them abandoned the study voluntarily. 1 left because she was pregnant, and 1 violated the protocol norms and was expelled.
Arm/Group | Less Oxidized Oil and Diet | More Oxidized Oil and Diet | Diet
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 3/20 | 0/18 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Less Oxidized Oil and Diet (N=20) | More Oxidized Oil and Diet (N=18) | Diet (N=19)
Violation of protocol norms (Investigations) | 0 | 0 | 1 — The participant did not follow the rules and the diet
Study abandonment (Social circumstances) | 3 | 0 | 0 — The participants lost interest in the diet and deciced to abandon the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No